CLINICAL TRIAL: NCT05060575
Title: The Effect of Education and Telephone Counseling Given to Hypertension Patients on Drug Medıcation Adherence and Rational Medication Use: Single-Blind Randomized Controlled Trial
Brief Title: Hypertension Patients on Drug Medication Adherence and Rational Medication Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Associate Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ayyuzlum3207
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Hypertension Patients
Keywords: Hypertension; Tele nursing; Education; Rational medication use; Drug medication adherence; Nursing
MeSH Terms: conditions — Hypertension | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDUTC (Experimental): Drug use and rational drug use training will be given to hypertension patients in the experimental group.
  The patients in the experimental group twice in the 1st month (2nd and 4th weeks), once in the 2nd month (8th week) and once in the 3rd month (12th week) phone call counseling will be providedved an average of 10-15 minutes.
  Interventions: Other: Education and Telephone Counceling
- Control Group (Active Comparator): Routine hospital care.
  Interventions: Other: Education and Telephone Counceling

INTERVENTIONS:
Other: Education and Telephone Counceling — Drug use and rational drug use training will be given to hypertension patients in the experimental group.
  The patients in the experimental group twice in the 1st month (2nd and 4th weeks), once in the 2nd month (8th week) and once in the 3rd month (12th week) phone call counseling will be providedved an average of 10-15 minutes.

SUMMARY:
This research will be conducted to determine the effects of education and telephone counseling given to hypertension patients on drug treatment compliance and rational drug use.

DETAILED DESCRIPTION:
This research will be conducted to determine the effects of education and telephone counseling given to hypertension patients on drug treatment compliance and rational drug use.

Research Hypotheses H0: Education and telephone counseling given to hypertension patients do not affect drug treatment compliance.

H1: Education and telephone counseling given to hypertension patients increase drug treatment compliance.

H0: Education and telephone counseling given to hypertension patients do not affect rational drug use.

H1: Education and telephone counseling given to hypertension patients increase rational drug use.

This study was planned as a single-blind randomized controlled experimental study.

ELIGIBILITY:
Inclusion Criteria:

* - Diagnosed with hypertension,
* Hypertension disease duration of at least 6 months,
* Using at least one drug due to hypertension,
* 18 years old and over
* Literate,
* Living in the town centre,
* Owns a phone
* Open to communication and cooperation,
* Patients willing to participate in the study will be included in the study.

Exclusion Criteria:

* Having a psychiatric illness
* Hearing loss,
* Can't understand or speak Turkish and
* Patients who do not wish to continue the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Adherence to Medication Self-Efficacy Scale | 12 weeks
  The scale consists of 13 items and determines the self-efficacy/confidence level of adherence to drug treatments of individuals with hypertension. The scale is evaluated by scoring from 1 to 4 in each question. The minimum score that can be obtained from the scale is 13, and the maximum score is 52. The increase in the scale score indicates that the compliance of individuals to antihypertensive drug treatment increases positively.
Rational Drug Use Scale | 12 weeks
  The scale has 36 items and is a triple Likert type. Behavioral beliefs (items 1-9), Control beliefs (items 10-16), Attitude (items 17-21), Subjective norm (items 22-23), Intention (items 24-28), and Knowledge It has 6 sub-dimensions (items between 29 and 36). Scoring of scale items was never (0), sometimes (1), and always (2) for positive items; negative items (items 13, 14, 17, 18, 19, 20, 21, and 24) are calculated as never (2), sometimes (1), and always (0). The scores that can be obtained from the scale range from 0 to 72. As the score obtained from the scale increases, the level of rational drug use increases.

SECONDARY OUTCOMES:
Diastolic/Systolic blood pressure | 12 weeks
  Systolic and Diastolic blood pressure will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GÖK UĞUR, Assoc., Principal Investigator — Ordu Ünivercity
Locations (1):
- Hacer GÖK UĞUR, Ordu, Cumhuriyet Campus Cumhuriyet District, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No